CLINICAL TRIAL: NCT02245776
Title: Autologous Bone Marrow Mononuclear Cell Therapy for Incurable Neurological Disorders
Brief Title: Stem Cell Therapy in Incurable Neurological Disorders
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-16
Record Dates: First submitted 2014-09-12; First posted 2014-09-22 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Neurological; Disorder, Nervous System
Keywords: Incurable Neurological Disorders; Autologous mononuclear cell therapy; Stem cells
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): Bone marrow mononuclear cell transplantation
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of the study was to analyze the benefit of autologous mononuclear cell therapy in incurable neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of incurable neurological disorders
* age above 6 months

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia
* pregnancy
* lactation

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in various clinical symptoms of neurological disorders | 1 year
  Change in various symptoms such as muscle strength, limb strength, ambulation, neck holding, bladder bowel management, spasticity, sensation, speech, etc depending on the disorder will be recorded at 1 year follow up. Percentage analysis of each symptom will be carried out to study the benefits of stem cell therapy on them.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No